CLINICAL TRIAL: NCT01006174
Title: Dietary Lipids as Primary Modulators of Carotenoid Absorption in Vegetables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph.D., Purdue University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0707005641
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Absorption of Carotenoids From Vegetables
MeSH Terms: interventions — Soybean Oil; Rapeseed Oil; Butter

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A (Experimental): Subjects will be assigned to consume 3 grams soybean oil, 8 grams canola oil, and 20 grams butter that is added to a salad.
  Interventions: Other: Soybean Oil; Other: Canola Oil; Other: Butter
- B (Experimental): Subjects will be assigned to consume 8 grams soybean oil, 20 grams canola oil, and 3 grams butter that is added to a salad.
  Interventions: Other: Soybean Oil; Other: Canola Oil; Other: Butter
- C (Experimental): Subjects will be assigned to consume 20 grams soybean oil, 3 grams canola oil, and 8 grams butter that is added to a salad.
  Interventions: Other: Soybean Oil; Other: Canola Oil; Other: Butter

INTERVENTIONS:
Other: Soybean Oil — Depending on the experimental group assigned, each subject which will be given one of three different amounts of soybean oil that is added to a salad.
Other: Canola Oil — Depending on the experimental group assigned, each subject which will be given one of three different amounts of canola oil that is added to a salad.
Other: Butter — Depending on the experimental group assigned, each subject which will be given one of three different amounts of butter that is added to a salad.

SUMMARY:
The purpose of this research study is to determine how dietary fats and oils influence the absorption of beneficial plant pigments (carotenoids) from vegetables. The study will examine changes in blood carotenoids in response to eating a salad with different fats/oils.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-50 years.
* Body mass index (BMI: weight (kg)/height (m2)) ranging from 20-29 kg/m²
* Weight stable (<4.5 kg change within the last 3 months),
* Constant habitual activity pattern, not to exceed activities of a recreational level over the past 3 months.
* Must be pre-menopausal
* Have clinically normal blood profiles (specifically normal liver and kidney functions and fasting blood glucose of ≤110 mg/dl)
* Non-smoking
* Non-diabetic
* No current or planned pregnancy
* Not using any hormone-based contraceptive, e.g., pill, patch, injection, implants, etc.
* No current use of medication affecting lipid profile
* No intestinal disorders including lipid malabsorption, lactose intolerance
* No heavy consumption of alcohol (>2 drinks per day)
* No current use of dietary supplements that affect cholesterol, (e.g. Benocol or fiber supplements) or a willingness to discontinue their use during the study.

Exclusion Criteria:

* Menopausal
* Diabetic
* Currently pregnant
* Currently using any type of hormone-based contraceptives, (e.g., pill, patch, injection, implants, etc.)
* Use of lipid altering medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Evaluating the impact of dietary lipid profiles on intestinal absorption of carotenoids from vegetables. | 66 days

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States